CLINICAL TRIAL: NCT01335191
Title: Clinical Study of TUTI-16 in Asymptomatic, HIV-1 Infected Subjects Effectively Controlled by Antiretroviral Therapy and the Effects on Viral Load During a Structured Treatment Interruption
Brief Title: Clinical Study of TUTI-16 in Asymptomatic HIV-1 Infected Subjects (THYMON-11001)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thymon, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THYMON-11001
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infections
Keywords: HIV; vaccine; lipopeptide; Tat; TUTI-16; THYMON
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TUTI-16 (1.0 mg) (Experimental): Two subcutaneous injections of 1.0 mg at Day 0 and Week 3.
  Interventions: Biological: TUTI-16 (1.0 mg)
- Placebo (Placebo Comparator): Two subcutaneous injections of placebo at Day 0 and Week 3.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TUTI-16 (1.0 mg) — Two subcutaneous injections of TUTI-16 (1.0 mg) at Day 0 and Week 3.
  Arms: TUTI-16 (1.0 mg)
Other: Placebo — Two subcutaneous injections of Placebo at Day 0 and Week 3.
  Arms: Placebo

SUMMARY:
This protocol represents the third in human study of TUTI-16, and is being conducted to gather additional safety and human immunogenicity (anti-HIV-1 Tat titers) data of subcutaneously administered TUTI-16.

DETAILED DESCRIPTION:
In this study, HIV-1 infected subjects on ART, with undetectable HIV-1 viral load, will be immunized with 1mg TUTI-16 or placebo in a randomized double blind fashion (prime and 3 week boost). Three weeks after the 3 week boost (week 6) ART will be stopped. HIV-1 viral load and CD4+ T-cell levels will be determined at defined intervals through 54 weeks (48 weeks Post ART discontinuation).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age ≥ 18 and ≤ 50 years at Screening
* Body weight of 50-100 kg (inclusive) at Screening.
* HIV-1 seropositive subjects on effective ART for > 12 months (undetectable HIV plasma viremia), viral set point before ART > 10,000.
* CD4+ T-cell count ≥ 500/mm3.
* No antiviral drug within 8 weeks of screening. Patients stabilized on Aciclovir and Valciclovir for more than 6 months may be enrolled.
* Karnofsky performance status > 90% at screening.
* In good health as determined by medical history, a baseline physical examination, vital signs, and clinical laboratory tests.
* Subject is willing and able to sign written informed consent prior to beginning study procedures.
* Subject is willing and able to follow instructions, comply with the protocol requirements and make all required study visits.

Exclusion Criteria:

* Females planning to become pregnant during the course of the study.
* Females with a positive pregnancy test at Screening or study enrollment.
* Any out-of range laboratory value at screening that has not been reviewed, approved and documented as not clinically significant by the Principal Investigator.
* Systemic infection or other vaccination within 6 weeks prior to screening. Live vaccine within 1 year of screening.
* Autoimmune disease (e.g., psoriasis, rheumatoid arthritis, etc.) or inflammatory bowel disease confirmed by clinical history.
* Positive at screen for HBV (by HBsAg assay) or HCV (by antibody ELISA) unless there is no active infection as judged by an elevated alanine aminotransferase (ALT) at screening.
* Alanine aminotransferase (ALT) above the upper limit of normal at screening.
* Hemoglobin outside of laboratory normal range at screening.
* Absolute neutrophil counts outside of laboratory normal range at screening.
* Platelet count outside of laboratory normal range at screening.
* A history of significant drug allergy.
* A general medical or psychological condition or behavior, including current substance dependence or abuse that, in the opinion of the investigator, might not permit the subject to complete the study or sign the informed consent.
* Subjects experiencing an acute Herpetic event.
* Any other condition or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening that, in the opinion of the Principal Investigator would make the subject unsuitable for the study or put them at additional risk.
* Routine or PRN consumption of immune suppressive medications that the subject is unable or unwilling to discontinue during the study.
* Inability to understand or follow study instructions.
* Participation in another investigational drug/vaccine study within 30 days preceding the first injection of investigational agent in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mardik Donikyan, MD, Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs, New York, New York, United States

REFERENCES:
- [Derived] Goldstein G, Damiano E, Donikyan M, Pasha M, Beckwith E, Chicca J. HIV-1 Tat B-cell epitope vaccination was ineffectual in preventing viral rebound after ART cessation: HIV rebound with current ART appears to be due to infection with new endogenous founder virus and not to resurgence of pre-existing Tat-dependent viremia. Hum Vaccin Immunother. 2012 Oct;8(10):1425-30. doi: 10.4161/hv.21616. Epub 2012 Oct 1. PMID 23095869

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TUTI-16 (1.0 mg) | Placebo
Started | 16 | 11
Completed | 16 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TUTI-16 (1.0 mg) | Placebo | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Customized [Mean (Full Range); unit: years]
  Between 18 and 65 years | 45 [27 to 55] | 43 [24 to 54] | 43 [24 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 14
  Male | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  United States | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Anti-Tat Antibody Titer
Description: ELISA based chemiluminescent assay to determine the anti-Tat antibody response
Time Frame: 54 weeks
Population: all subjects enrolled
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | TUTI-16 (1.0 mg) | Placebo
Number analyzed (Participants) | 16 | 11
ng/mL | 698 [0 to 3000] | 4 [0 to 42]

ADVERSE EVENTS:
Arm/Group | TUTI-16 (1.0 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 8/16 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TUTI-16 (1.0 mg) (N=16) | Placebo (N=11)
injection site reaction (General disorders) | 8 (13) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No